CLINICAL TRIAL: NCT03564236
Title: Nasal High-Flow Therapy to Treat COPD Exacerbations: a Matter of Monitoring and Controlling Settings?
Brief Title: Nasal High-Flow in COPD
Acronym: High-TeC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marieke Duiverman (Other)
Collaborators: Rijnstate Hospital (Other); Medisch Spectrum Twente (Other); Albert Schweitzer Hospital (Other); Technical University of Twente (Other); Fisher and Paykel Healthcare (Industry); Vivisol (Other)
Responsible Party: Sponsor-Investigator, Marieke Duiverman, Principal Investigator, University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201800398
Record Dates: First submitted 2018-05-23; First posted 2018-06-20 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: COPD Exacerbation
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Paralell-group randomised controlled trial
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Active Comparator): Standard care is provided according to our local COPD exacerbation protocol. All patients are treated with:
  * oral prednisolone 40 mg/day for 5 days;
  * antibiotics prescribed according to the following criteria: fever (body temperature > 38.5 degrees Celsius), elevated C-reactive protein (CRP) >50, change in sputum colour, and/or according to the physician's decision of severe illness, and/or in all patients with a FEV1 <30% of predicted;
  * high dose inhaled corticosteroids, beta-agonists and or anticholinergics.
  * Oxygen will be prescribed in all patients through a standard low flow system in order to maintain an adequate arterial oxygen saturation (Sa,O2) Patients will be discharged with regular low flow oxygen once they fulfil the criteria for long-term oxygen therapy.
  Interventions: Other: Standard care
- Nasal High Flow Therapy (Experimental): In addition to the standard care described above, patients in the intervention group will be treated with:
  * nHFT, set at 30-50 L/min flow with oxygen to achieve an adequate oxygen saturation. nHFT is prescribed for at least 6 hours, but patients are stimulated to use the device as much as possible during the hospital stay.
  * During periods without HFT through a standard low flow system, to maintain an adequate arterial oxygen saturation (Sa,O2) (between 90-92% if patients are concomitantly hypercapnic, and between 90-95% if patients are normocapnic). Flow rates are titrated accordingly.
  * After discharge patients in the nHFT arm will continue the prescribed therapy at home for 90 subsequent days.
  Interventions: Device: Nasal High Flow Therapy

INTERVENTIONS:
Device: Nasal High Flow Therapy — Nasal High Flow Therapy (nHFT) is an innovative therapy for patients with respiratory diseases. It supplies heated, humidified, and oxygen-enriched air at high flow rates through a nasal cannula. Because the air is provided through an open system with a nasal cannula, it is relatively easy to apply and suggested to be very comfortable for patients. The technique has been shown to be effective in the treatment of hypoxemic respiratory failure, mainly in neonates[2] and patients with acute hypoxemic respiratory failure on intensive care units (ICU).[3]
  Arms: Nasal High Flow Therapy
Other: Standard care — Standard regular care of a COPD exacerbation
  Arms: Standard Care

SUMMARY:
Rationale: Chronic Obstructive Pulmonary Disease (COPD) is a disease with high morbidity and mortality worldwide. COPD exacerbations are the important contributor to disease deterioration and decrease in health-related quality of life (HRQoL). Since therapeutic options to treat exacerbations effectively are limited, many patients have persistent loss of vital functioning and suffer from frequent re-hospitalisations.

Nasal high flow therapy (nHFT) is an innovative therapy that provides humidified and heated air through a nasal cannula. Although there is some preliminary evidence that nHFT is effective in stable COPD patients, there are no data at all regarding the effectiveness of nHFT in COPD exacerbations. A key problem in the implementation of nHFT is that the underlying working mechanisms are not clear and therefore the appropriate way to apply nHFT is unknown.

Objective: The aim of the present study is to prove efficacy of nHFT in enhancing recovery from COPD exacerbations. We aim to improve the effectiveness of nHFT by developing new technologies to control and monitor the effect of nHFT and by providing background for optimal settings of nHFT.

Study design: The study will be designed as a multicentre randomised controlled trial, with the University Medical Center Groningen, the "Medisch Spectrum Twente", "Albert Schweizer ziekenhuis", Rijnstate hospital, and the University of Twente, collaborating.

Study population: One hundred thirty-six patients with known COPD GOLD stage II to IV and hypoxemic respiratory failure hospitalised with a COPD exacerbation will be included.

Intervention (if applicable): Patients will be randomised to standard care or nHFT (≥ 6 hours/day) during hospitalisation and the 90 days after discharge, as added to standard care.

Main study parameters/endpoints: The primary outcome will be improvement in HRQoL after 90 days.

DETAILED DESCRIPTION:
The study will be a parallel group 2-arms non blinded multicentre 2-phase randomised controlled trial comparing the effect of nHFT on subjective recovery in COPD patients admitted to the hospital for a COPD exacerbation as compared to the standard care. First, we will define the optimal setting and gain more insight in insight in mechanisms why and how nHFT might work in a subpopulation, then continuing with inclusion in the randomized controlled trial including the 136 patients in total to prove efficacy in terms of patient-centered outcomes. To get more insight in mechanisms why and how nHFT might work we incorporate: a) neuromechanical investigations and analyses; and b) anatomical investigations, both in patients and in experimental models, the latter in order to minimise patient effort.

ELIGIBILITY:
Inclusion Criteria:

Patients have to fulfil all of the following inclusion criteria:

* History of COPD Global Initiative of Obstructive Lung Diseases (GOLD) stage II to IV (FEV1< 80% of predicted with an FEV1/forced vital capacity (FVC) ratio <70), with a history of at least 10 pack years smoking.
* Being admitted to the hospital with a COPD exacerbation
* Signs of compensated respiratory failure (hypercapnia (partial arterial carbon dioxide pressure (PaCO2) ≥ 6.0 kPa and/or hypoxemia (partial arterial oxygen pressure (PaO2) ≤ 8.0 kPa at room air), with pH > 7.34
* At least 2 COPD exacerbations in the year prior to the index hospital admission (exacerbation defined as worsening of pulmonary symptoms requiring oral steroids and/or antibiotics and/or hospital admission)
* Written informed consent is obtained

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* No lung function data available
* The presence of another acute condition (e.g. pneumonia, acute congestive heart failure, pulmonary embolus) explaining or significantly contributing to the index admission
* Inability to comply with the tests
* The presence of another chronic lung disease (e.g. asthma, restrictive lung disease).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life | 90 days
  The primary outcome will be improvement in HRQoL, defined as the net response rate on the St. George Respiratory questionnaire (SGRQ) after 90 days

SECONDARY OUTCOMES:
Treatment failure | 90 days, follow-up up to 1 year
  Treatment failure of nHFT, defined as death, need for intensive care admission for respiratory failure, need for (non)-invasive mechanical ventilation, during the study period, in patients randomised to nHFT.
Hospitalisations | 90 days, follow-up up to 1 year
  Hospital length of stay of the index admission, readmissions, readmission characteristics and complications.
Exacerbation frequency | 90 days, follow-up up to 1 year
  Exacerbations will be defined as periods of symptom worsening treated with oral prednisolone and/or antibiotics.
Severe Respiratory Insufficiency Questionnaire (SRI) | 90 days
  Subjective recovery during hospitalisation and thereafter will also be investigated by assessing the Severe Respiratory Insufficiency Questionnaire (SRI). This is a well-known and validated Health-Related quality of Life (HRQoL) questionnaire especially designed for patients with chronic hypercapnic respiratory failure containing 49 items measuring 7 conceptual domains of HRQoL: respiratory complaints, physical functioning, attendant symptoms and sleep, social relationships, anxiety, psychological well-being and social functioning, and a summary score. The domain scores are calculated by transforming the mean item score into a percentage ranging from 0 (most severely depressed health status as complaints/limitations are severe) to 100 (perfect health status with no complaints/limitations).
Clinical COPD Questionnaire (CCQ) | 90 days
  Subjective recovery during hospitalisation and thereafter will be also investigated by assessing the Clinical COPD Questionnaire (CCQ). The CCQ is a disease specific but not "respiratory failure" specific questionnaire. It is a 10-item, self-administered questionnaire that can be completed in less than 2 minutes, and as so, is an attractive measure to be performed repeatedly during an exacerbation. Items are divided into three domains: symptom, functional state and mental state; patients are required to respond to each item on a seven-point Likert scale where 0 = asymptomatic/no limitation and 6 = extremely symptomatic/total limitation. The final score is the mean of all ten items, and scores for the three domains can be calculated separately if required.
Euroqual-5 Dimensions questionnaire (EQ-5D) | 90 days
  Subjective recovery during hospitalisation and thereafter will also be investigated by assessing the EQ-5D. The EQ-5D questionnaire is made up for two components; health state description and evaluation. In description part, health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The respondents self-rate their level of severity for each dimension using five-level (EQ-5D-5L) scale.
  In evaluation part, the respondents evaluate their overall health status using the visual analogue scale (EQ-VAS), ranging from 0 to 100.
  EQ-5D-5L health states, defined by the EQ-5D-5L descriptive system, will be converted in index values, facilitating the calculation of quality-adjusted life years (QALYs) that are used to inform economic evaluations of health care interventions, according to the guideline (https://euroqol.org).
Cough and Sputum Assessment Questionnaire (CASA-Q) | 90 days
  Subjective recovery during hospitalisation and thereafter will also be investigated by assessing the Cough and Sputum Assessment Questionnaire (CASA-Q). CASA-Q score is a tool for evaluating cough and sputum and their impact on patient's QOL in COPD. CASA-Q consists of two cough domains; the cough symptom domain (COUS, 11 items) and the cough impact domain (COUI, 8 items), and two sputum domains; the sputum symptom domain (SPUS, 3 items) and the sputum impact domain (SPUI, 16 items). All items will be scored from 0 to 4, such that the score was 0-12 for COUS and SPUS, and 0 to 24 for SPUI, and 0 to 32 for COUI, and each item summed and rescaled using the following algorithm: (sum rescored items)/(range of rescored item sum) x 100 (%). This results in CASA-Q scores that range from 0 to 100, with higher score associated with fewer symptoms and less impact due to cough and sputum.
Gas exchange | 90 days
  Gas exchange will be monitored with both arterial blood gases during spontaneous breathing at daytime and nocturnal transcutaneous monitoring while on the prescribed therapy.
Functional capacity | discharge and after 90 days
  Functional capacity will be assessed at discharge and 90 days thereafter (T1 and T3) by means of calculating daily activity level, measured with a step counter
Assessment of cardiac function | 90 days
  An electrocardiogram (ECG) and blood pressure measurements will be performed. The N-terminal of the brain natriuretic peptide (NTproBNP) will be assessed by routine laboratory methods.
Compliance | 90 days
  Compliance with the nHFT device will be read out from the compliance logs stored in the device when patients visit the outpatient clinic.
Cost-effectiveness | 90 days
  Cost-effectiveness will be investigated by estimating the healthcare costs of nHFT and usual care and the HRQoL gains of usual care and nHFT.

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Rijnstate Hospital, Arnhem
  - Albert Schweizer ziekenhuis, Dordrecht
  - University Medical Center Groningen, Groningen

IPD SHARING:
Plan to Share IPD: Undecided